CLINICAL TRIAL: NCT04318522
Title: Effect of Conventional Transcranial Direct Current Stimulation (c-tDCS) and High-definition Transcranial Direct Current Stimulation (HD-tDCS) on the Prefrontal Cortex
Brief Title: Non-Invasive Brain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Chairman and Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017.331
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation Group (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulator
- Control Group (Sham Comparator)
  Interventions: Device: Transcranial Direct Current Stimulator

INTERVENTIONS:
Device: Transcranial Direct Current Stimulator — Transcranial Direct Current Stimulation (tDCS) is a non-invasive brain stimulation device that can excite or inhibit the brain activity depending on the stimulation protocol. It has mainly two variants including conventional c-tDCS and High-Definition HD-tDCS.

SUMMARY:
The study focusses on utilizing neuroimaging modalities, including Electroencephalography (EEG) and Functional Magnetic Resonance Imaging (fMRI) to study the impact of non-invasive brain stimulation on the prefrontal cortex during a cognitive task.

DETAILED DESCRIPTION:
In this study, a total of 40 subjects will be randomly assigned to 2 groups i.e. experimental and sham. Conventional transcranial direct current stimulation (c-tDCS) and high-definition transcranial direct current stimulation (HD-tDCS) will be used to stimulate the prefrontal cortex of the brain. EEG and fMRI will be collected before, during and after stimulation to understand the impact of stimulation on brain dynamics. The investigators hypothesize that the stimulation of the prefrontal cortex will improve performance during cognitive tasks along with changes in the neural processing detected by neuroimaging modalities.

ELIGIBILITY:
Inclusion Criteria:

* Right Handedness,
* Age > 18

Exclusion Criteria:

* History of any other neurological disease,
* Any psychological or psychiatric disease,
* Significant visual or auditory impairments,
* tDCS contraindications including implanted metallic or electronic devices, seizures or convulsions, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Reaction Time (RT) | 1 hour
  Reaction time of the subject during a cognitive task would be a measure to assess changes in performance due to stimulation
Concentration Rate | 1 hour
  The percentage of accurate responses during the cognitive task within the stipulated time will be calculated to see an impact on concentration after stimulation
Event related potential latency and amplitude | 1 hour
  Changes in latency and amplitude of event related potentials including P300 & N200 would be used as neural marker to understand cognitive processing in the brain.
Functional Magnetic Resonance Imaging (fMRI) | 1 hour
  Changes in fMRI connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan A, Chen C, Eden CH, Yuan K, Tse CY, Lou W, Tong KY. Impact of anodal high-definition transcranial direct current stimulation of medial prefrontal cortex on stroop task performance and its electrophysiological correlates. A pilot study. Neurosci Res. 2022 Aug;181:46-54. doi: 10.1016/j.neures.2022.03.006. Epub 2022 Apr 1. PMID 35378119
- [Derived] Khan A, Wang X, Ti CHE, Tse CY, Tong KY. Anodal Transcranial Direct Current Stimulation of Anterior Cingulate Cortex Modulates Subcortical Brain Regions Resulting in Cognitive Enhancement. Front Hum Neurosci. 2020 Dec 16;14:584136. doi: 10.3389/fnhum.2020.584136. eCollection 2020. PMID 33390917